CLINICAL TRIAL: NCT05225376
Title: Physical Activity and Sedentary Lifestyle During Pregnancy: Feasibility and Impact Study on Sedentary Behavior
Acronym: PregMouv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2021 VENDITTELLI; 2021-A01683-38 (Other: 2021-A01683-38)
Record Dates: First submitted 2022-01-12; First posted 2022-02-04 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Sedentary Behavior; Pregnancy Related; Perinatal Problems; Sedentary Time; Morbidity;Perinatal
Keywords: pregancy; exercice; sedentary; maternal morbidity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: all participants will receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Establishment of physical activity sessions for pregnant women (Experimental): All the women will receive the studied intervention
  Interventions: Other: Physical activity sessions for pregnant women

INTERVENTIONS:
Other: Physical activity sessions for pregnant women — The physical activity sessions will take place once a week at the Estaing UHC, in the room used for the childbirth and parenting preparation classes of the outpatient obstetrics-gynecology clinic; and twice a week on Zoom. These sessions will be supervised by an APA professional (degree in STAPS and APA).
  The measurement of the women's physical conditions will make it possible to adapt and individualize the PA sessions to each woman's level.

SUMMARY:
Background:

Physical activity (PA) has beneficial effects on health, physical condition, and the maintenance of autonomy and independence at all ages of life. It also has numerous benefits during pregnancy: maintenance or improvement of physical condition, prevention of excessive weight gain, aid in postpartum weight loss, prevention of gestational hypertension, reduction in number of macrosomic infants at birth, reduction in lower back and pelvic pain, and prevention and improvement of postpartum depressive symptoms. A recent systematic review of the literature concluded that interventions to increase PA levels among pregnant women have a positive effect on this level. The studies included in the review also showed that these interventions have a positive effect on these women's well-being and their mental and physical health. Nonetheless, no study has examined this subject in France. Moreover, to our knowledge, no study in the international literature has looked at online interactive video sessions of PA during pregnancy.

Overall, few studies allow an assessment of the effect of sedentary behavior and inadequate PA during pregnancy on maternal, neonatal, or infant outcomes. This is equally true for the health of adults whose mothers were physically active during pregnancy. Moreover, we do not know the actual level of PA of women in France. Finally, we do not know what types of intervention described in the literature would enable the best adherence by French women to their initiation or maintenance of an adequate PA level.

Study hypothesis:

Our hypothesis is that setting up a free program of physical and sports activity session for pregnant women will enable them to meet the guidelines for PA practice during this period and to reduce their sedentary behavior.

Objectives:

1.1. Principal objective To study the feasibility of setting up physical activity (PA) sessions for pregnant women during their prenatal care, by assessing its acceptability, the perceived difficulty of the sessions, and their satisfaction with these sessions.

1.2. Secondary objectives

* To evaluate the effect of these sessions:

  * on the PA level and sedentary behavior of pregnant women,
  * on their quality of life (QoL).
* The feasibility and impact of the sessions will be studied according to their PA level at inclusion: active or inactive.
* To identify the facilitators of and obstacles to the acceptability of these sessions, other than those studied in the objectives above.
* To measure the willingness to pay of pregnant women so that we can quantify how much they would be willing to pay for such a program, were it were not free. Willingness to pay (measured in €) makes it possible to measure indirectly the acceptability of the program to the participants and the monetary value they attribute to it.

DETAILED DESCRIPTION:
Type of study:

Prospective interventional cohort feasibility study of PA sessions for pregnant women.

Number of centers: 1

One center: the Clermont-Ferrand university hospital center

Study description:

The study is based on voluntary participation in organized sessions of PA. For each woman the program will comprise 51 sessions (for a woman giving birth after 39 weeks of gestation) with three sessions a week starting between 21+6 d and 23+6 d weeks through 39+0 d weeks. Women will be asked to attend all three sessions each week. Each session will include a maximum of 5 women and will last for 45 minutes, with 30 minutes of endurance (aerobic) PA, as well as muscle (strength) training and some stretching. They will also include advice to women to limit their sedentary time and to allow them to perform PA outside of these sessions with an instructor. In addition to the mandatory weekly session in person, two sessions will be proposed as interactive video classes. A Zoom® link will be offered to the women so that they can connect to these two weekly sessions, taught by the adapted PA (APA) professional who teaches the in-person sessions. These sessions will have the same format as the in-person session (45 minutes) with viewing of both the APA professional (trainer/coach) and the participants (who can choose to be masked). The APA professional will also see the participants and thus can at any time correct their positions and give them individualized advice.

Study plan and procedures:

The women will be informed about the study from their first trimester of pregnancy. If they want to participate in the study and the PA sessions, they must contact the research midwife. Before their first participation in a PA session, each woman will meet with the research midwife, who will review with her the information about the study, verify the eligibility criteria, and obtain her written informed consent. During the first session, the woman will perform two physical ability tests (described below) with the APA instructor, to determine her initial PA level and her physical capacities.

At the end of each session, the instructor will record the women present or connected and evaluate the perceived difficulty of the session by having the women complete in their notebooks the Borg rating of perceived exertion, the scale of intensity according to the affective valence, and the conversation test.

At the end of the sixth month of gestation (28 weeks), the women will retake these physical ability tests with the instructor, complete the self-administered acceptability questionnaires and the PPAQ on line or in person. At the end of the eighth month of gestation (37 weeks), the women will retake these physical ability tests with the instructor, complete the self-administered acceptability questionnaires, and the PPAQ, on line or in person. At the end of their personnal program, the women will complete on line or in person the self-administered acceptability and satisfaction questionnaires and the WHOQOL-Brief. A short semi-directive telephone interview will then be performed to identify the facilitators of and obstacles to acceptability.

ELIGIBILITY:
Inclusion Criteria:

Adult pregnant women receiving prenatal care at the Estaing UHC maternity ward,

* Seen for prenatal care before the 21st week of gestation and booked to give birth at the Estaing UHC
* Agreeing to follow the full PA program proposed,
* Able to provide informed consent to participate in research,
* And covered by the national health insurance fund (or an affiliate).

Exclusion Criteria:

* Multiple pregnancy,
* With a relative or absolute contraindication to performing PA physical activity (see Tables 1 and 2, extracted from the French national authority for health guidelines for physical activity during pregnancy),
* Under guardianship or conservatorship,
* Or refusing to participate in the study.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Establishing Adherence of PA sessions during pregnancy | through study completion, an average of 1 year
  Women's adherence to the sessions proposed (% who attend all sessions until delivery).
Establishing perceived difficulty of PA sessions during pregnancy | through study completion, an average of 1 year
  The perceived difficulty of the sessions will be evaluated by the women themselves with a self-administered questionnaire.
Establishing women's satisfaction of PA sessions during pregnancy | day1
  Satisfaction with the PA sessions for pregnant women during their prenatal care will be based on a self-administered questionnaire. Women's overall satisfaction with the sessions will be assessed on a numeric scale ranging from 0 to 10.
Establishing women's satisfaction of PA sessions during pregnancy | day 70
  Satisfaction with the PA sessions for pregnant women during their prenatal care will be based on a self-administered questionnaire. Women's overall satisfaction with the sessions will be assessed on a numeric scale ranging from 0 to 10.
Establishing women's satisfaction of PA sessions during pregnancy | day 133
  Satisfaction with the PA sessions for pregnant women during their prenatal care will be based on a self-administered questionnaire. Women's overall satisfaction with the sessions will be assessed on a numeric scale ranging from 0 to 10.

SECONDARY OUTCOMES:
Pregnant women's PA level and sedentary behavior | before the first PA session, at the end of the sixth month of gestation, and at the end of all the sessions (9 months)
  These will be assessed with the French version of the PPAQ (Pregnancy Physical Activity Questionnaire) questionnaire. Their physical condition will also be assessed by physical ability tests (Cardiopulmonary endurance (6-minute walk test); Handgrip test with dynamometer) , all conducted by the APA instructors.
Changes in these pregnant women's quality of life | Before the first PA session, at 6 months of gestation, and at the end of all the sessions (9 months)
  The pregnant women's QoL will be assessed with the self-administered WHOQOL-Brief questionnaire, which has been validated in French. It was chosen because it specifically evaluates comprehensive/overall QoL over the past 2 weeks. It is a generic, multidimensional questionnaire. It explores 6 dimensions (physical health, psychological well-being, satisfaction with life, social relationships, environment, and spirituality). A score is calculated from each item. A user manual is available, free of charge, from the WHO web site.
The facilitators of and obstacles to the sessions' acceptability will be assessed in semi-directive interviews conducted by a midwife. | at the end of all the sessions (9 months)
  These interviews, based on a semi-directive interview guide, will focus on the following themes: (1) the perceived importance of PA during pregnancy; (2) the level of understanding and appropriation of the support procedures provided during the pregnancy; (3) satisfaction with the workshops proposed and their relation with daily QoL; (4) suggestions for improvement to better meet women's expectations. The estimated duration of these interviews is from 30 to 45 minutes.
Willingness to pay | at the end of all the sessions (9 months)
  This will be collected during the interview. The pregnant women will be asked how much they would be willing to pay to participate in such a program, outside of the study. If the willingness to pay is low, the interviewer can then organize the discussion around the financial obstacles: nonreimbursement by health insurance, economic situation, and nonadherence.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Vendittelli, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haute Autorité de Santé. Guide de promotion, consultation et prescription médicale d'activité physique et sportive pour la santé chez les adultes [Internet]. 2019. Disponible sur: https://www.has-sante.fr/upload/docs/application/pdf/2018-10/guide_aps_vf.pdf
- [Background] Institut national de la santé et de la recherche médicale (France). Activité physique: prévention et traitement des maladies chroniques. 2019.
- [Background] Organisation mondiale de la santé. Recommandations mondiales sur l'activité physique pour la santé. Genève: OMS; 2010.
- [Background] Haute Autorité de Santé. Prescription d'activité physique et sportive Pendant la grossesse et en post-partum [Internet]. Saint-Denis: HAS; [cité 2 mars 2020] p. 14. Disponible sur: https://www.has-sante.fr/upload/docs/application/pdf/2019-07/app_329_ref_aps_grossesse_vf.pdf
- [Background] Agence nationale de sécurité sanitaire, de l'alimentation, de l'environnement, et du travail. Actualisation des repères du PNNS - Révisions des repères relatifs à l'activité physique et à la sédentarité [Internet]. Maison-Alfort; 2016 [cité 15 juill 2020]. Disponible sur: https://www.anses.fr/fr/system/files/NUT2012SA0155Ra.pdf
- [Background] Verdot C, Salanave B, Deschamps V. Activité physique et sédentarité dans la population française. Situation en 2014- 2016 et évolution depuis 2006-2007. Bull Epidémiol Hebd. 2020;15:296-304.
- [Background] Équipe de surveillance et d'épidémiologie nutritionnelle (Esen). Étude de santé sur l'environnement, la biosurveillance, l'activité physique et la nutrition (Esteban), 2014-2016. Volet Nutrition. Chapitre Activité physique et sédentarité. 2e édition [Internet]. Saint-Maurice: Santé publique France; 2020 p. 58. Disponible sur: www.santepubliquefrance.fr
- [Background] DIVISION OF MENTAL HEALTH AND PREVENTION OF SUBSTANCE ABUSE WORLD HEALTH ORGANIZATION. WHOQOL User Manual [Internet]. WHO; 2012 [cité 21 oct 2020] p. 106. Disponible sur: https://apps.who.int/iris/bitstream/handle/10665/77932/WHO_HIS_HSI_Rev.2012.03_eng.pdf?sequence=1&isAllowed=y
- [Background] Inserm (dir.). Activité physique : contextes et effets sur la santé. Rapport. [Internet]. Les éditions Inserm. Paris; 2008 [cité 23 juill 2020]. 811 p. Disponible sur: http://www.ipubli.inserm.fr/bitstream/handle/10608/97/expcol_2008_activite.pdf?sequence=1
- [Result] Ekelund U, Tarp J, Steene-Johannessen J, Hansen BH, Jefferis B, Fagerland MW, Whincup P, Diaz KM, Hooker SP, Chernofsky A, Larson MG, Spartano N, Vasan RS, Dohrn IM, Hagstromer M, Edwardson C, Yates T, Shiroma E, Anderssen SA, Lee IM. Dose-response associations between accelerometry measured physical activity and sedentary time and all cause mortality: systematic review and harmonised meta-analysis. BMJ. 2019 Aug 21;366:l4570. doi: 10.1136/bmj.l4570. PMID 31434697
- [Result] Fazzi C, Saunders DH, Linton K, Norman JE, Reynolds RM. Sedentary behaviours during pregnancy: a systematic review. Int J Behav Nutr Phys Act. 2017 Mar 16;14(1):32. doi: 10.1186/s12966-017-0485-z. PMID 28298219
- [Result] Brekke I, Richardsen KR, Jenum AK. Sickness absence in pregnancy and sedentary behavior: a population-based cohort study from Norway. BMC Public Health. 2019 Jan 16;19(1):71. doi: 10.1186/s12889-018-6379-4. PMID 30651106
- [Result] Barone Gibbs B, Paley JL, Jones MA, Whitaker KM, Connolly CP, Catov JM. Validity of self-reported and objectively measured sedentary behavior in pregnancy. BMC Pregnancy Childbirth. 2020 Feb 11;20(1):99. doi: 10.1186/s12884-020-2771-z. PMID 32046663
- [Result] van der Waerden J, Nakamura A, Pryor L, Charles MA, El-Khoury F, Dargent-Molina P; EDEN Mother-Child Cohort Study Group. Domain-specific physical activity and sedentary behavior during pregnancy and postpartum depression risk in the French EDEN and ELFE cohorts. Prev Med. 2019 Apr;121:33-39. doi: 10.1016/j.ypmed.2019.02.012. Epub 2019 Feb 11. PMID 30763624
- [Result] Poudevigne MS, O'Connor PJ. A review of physical activity patterns in pregnant women and their relationship to psychological health. Sports Med. 2006;36(1):19-38. doi: 10.2165/00007256-200636010-00003. PMID 16445309
- [Result] Chan CWH, Au Yeung E, Law BMH. Effectiveness of Physical Activity Interventions on Pregnancy-Related Outcomes among Pregnant Women: A Systematic Review. Int J Environ Res Public Health. 2019 May 23;16(10):1840. doi: 10.3390/ijerph16101840. PMID 31126153
- [Result] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Result] Teychenne M, Abbott G, Stephens LD, Opie RS, Olander EK, Brennan L, van der Pligt P, Apostolopoulos M, Ball K. Mums on the Move: A pilot randomised controlled trial of a home-based physical activity intervention for mothers at risk of postnatal depression. Midwifery. 2021 Feb;93:102898. doi: 10.1016/j.midw.2020.102898. Epub 2020 Nov 27. PMID 33290891
- [Result] Chandonnet N, Saey D, Almeras N, Marc I. French Pregnancy Physical Activity Questionnaire compared with an accelerometer cut point to classify physical activity among pregnant obese women. PLoS One. 2012;7(6):e38818. doi: 10.1371/journal.pone.0038818. Epub 2012 Jun 11. PMID 22701717
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Arcuri JF, Borghi-Silva A, Labadessa IG, Sentanin AC, Candolo C, Pires Di Lorenzo VA. Validity and Reliability of the 6-Minute Step Test in Healthy Individuals: A Cross-sectional Study. Clin J Sport Med. 2016 Jan;26(1):69-75. doi: 10.1097/JSM.0000000000000190. PMID 25706661
- [Result] Baumann C, Erpelding ML, Regat S, Collin JF, Briancon S. The WHOQOL-BREF questionnaire: French adult population norms for the physical health, psychological health and social relationship dimensions. Rev Epidemiol Sante Publique. 2010 Feb;58(1):33-9. doi: 10.1016/j.respe.2009.10.009. Epub 2010 Jan 21. PMID 20096515